CLINICAL TRIAL: NCT01956435
Title: Excimer Light Treatment for Idiopathic Guttate Hypomelanosis: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Collaborators: American Society of Dermatologic Surgeons (Unknown); Photomedex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR-13-151
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Idiopathic Guttate Hypomelanosis
MeSH Terms: interventions — Lasers, Excimer; Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Excimer Light Treatment Right Leg, Control Left Leg (Other): Excimer light treatment will be performed on the right leg of every subject, no treatment on the left or control leg of the subject.
  Interventions: Device: Excimer Light Treatment
- Excimer Light Treatment Left Leg, Control Right Leg (Other): Excimer light treatment will be performed on the left leg of every subject, no treatment on the right or control leg of the subject.
  Interventions: Device: Excimer Light Treatment

INTERVENTIONS:
Device: Excimer Light Treatment — Excimer light treatment will be performed on one leg of every subject as the intervention while the subjects other leg will serve as a control
  Other Names: Xtrac; Excimer laser; phototherapy

SUMMARY:
This pilot study will consist of 10 adult subjects with symmetric idiopathic guttate hypomelanosis on the lower legs. Subjects will be randomized to which extremity (right or left) will be treated. Treatments with the Xtrac Excimer laser will be performed twice weekly for 12 weeks using the typical vitiligo protocol. Our goal is to determine the effectiveness of excimer laser for repigmentation of idiopathic guttate hypomelanosis. Effectiveness will be graded by the blinded observer scale via photographic comparisons and will be graded by subject via survey every 4 weeks.

DETAILED DESCRIPTION:
Methods: This pilot study will consist of 10 adult subjects with symmetric IGH on the lower legs. After enrollment, 5 lesions of IGH on each leg will be selected by either Dr. Jennifer Gordon or Dr. Ammar Ahmed and marked. Subjects will be randomized to which extremity (right or left) will be treated. Treatments with the Xtrac Excimer laser (wavelength of 308nm) will be performed twice weekly for 12 weeks using the typical vitiligo protocol (see Appendix C). Photographs of both extremities will be taken prior to initial treatment and then every 4 weeks. The photographs will be analyzed by two separate, blinded dermatologists and rated on improvement from baseline using the following scale: 1= worsening of IGH; 2= no improvement (IGH remained stable); 3= mild improvement of IGH (some repigmentation on <50% IGH); 4= moderate improvement (some repigmentation on >50% or full repigmentation on <75% IGH); 5= full repigmentation on >75% IGH (see Appendix A). Subjects will also be asked to complete this survey subjectively every 4 weeks. Internal control will be represented by the marked lesions on the non-treated extremity of each patient. Control versus treatment groups will be statistically compared; however, due to the limited number of patient in this pilot study, a descriptive trend analysis will likely be completed. Subjects will be compensated $10 per visit (totaling $250). If a subject withdraws early from the study, they will be compensated for every completed visit. The 25th visit will consist of final photographs and surveys, and will not include treatment.

Statistical Analysis: The main outcomes to be collected are the improvement of IGH from baseline at weeks 4, 8 and 12 by the blinded dermatologists and by the subjects. Subjects will be stratified by Fitzpatrick skin type for analysis as well.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of idiopathic guttate hypomelanosis on the bilateral lower extremities with at least 5 lesions on each leg that are overall symmetric as determined by study personnel
* Patients must be 18 years or older
* Patients may be from any ethnicity but are required to be English-speakers
* Patients must provide written informed consent to participate in the study

Exclusion Criteria

* Patients with pre-existing dermatological condition that is exacerbated by ultraviolet radiation
* Non-English speakers
* Patients taking medications known to have potential phototoxic reactions
* Use of Ultraviolet tanning beds, Ultraviolet-A, Ultraviolet- B or excimer therapy within the previous 3 months on the lower extremities
* Current or previous treatment within the past 3 months specifically for IGH
* Pregnancy or pregnancy within the past 3 months (this can cause changes in pigmentation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Ahmed, MD, Principal Investigator — Seton Healthcare Family
Locations (1):
- Seton Family of Hospitals- Trinity Clinic, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Excimer Light Treatment Right Leg, Control Left Leg: Excimer light treatment will be performed on patients randomized to receive treatment on the right leg and left leg will be untreated control
- Excimer Light Treatment Left Leg, Control Right Leg: Excimer light treatment will be performed on patients randomized to receive treatment on the left leg and right leg will be untreated control
Period: Overall Study
Arm/Group | Excimer Light Treatment Right Leg, Control Left Leg | Excimer Light Treatment Left Leg, Control Right Leg
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This pilot study included six patients with idiopathic guttate hypomelanosis on their lower extremities, which were recruited from an outpatient dermatology clinic.
Groups:
- All Participants: All Study Participants
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Outcome
Description: Effectiveness will be graded by the blinded observer scal via photographic comparisons at the end of the study. Efficacy was assessed by improvement from baseline using the following scale: -1 = Worsening of IGH; 0 = No Improvement (IGH remained stable); 1 = Mild improvement of IGH (some re-pigmentation on <50% IGH); 2 = Moderate improvement (some re-pigmentation on >50% or full re-pigmentation on <75% IGH); 3 = Full re-pigmentation on >75% IGH.
Time Frame: 12 weeks
Population: healthy adult patients with bilateral IGH lesions on lower extremities
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Excimer Light Treatment: Lesions treated with excimer light
- Control: Lesions not treated with excimer light
Arm/Group | Excimer Light Treatment | Control
Number analyzed (Participants) | 6 | 6
units on a scale | 2.31 [2.08 to 2.54] | 1.15 [0.92 to 1.39]

2. Secondary Outcome: Subject Self-reported Assessment of Re-pigmentation for Treated Lesions
Description: Subject reported level of re-pigmentation for treated lesions was assessed by improvement from baseline using a scale from 1 - 4 with 1 being the least amount of re-pigmentation and 4 being the most re-pigmentation: 1 = Worsening of the light spots that were treated (the light spots seem to have gotten lighter or I have more light spots in the areas that were treated); 2 = No Improvement of the light spots (light spots have not changed since starting this study); 3 = Mild improvement of the light spots (there is some darkening of the light spots, but not in more than half of them); 4 = Moderate improvement (there is some darkening of the light spots in more than half of the light spots, but not more than 75% of them).
Time Frame: 12 weeks
Population: healthy adult patients with bilateral IGH lesions on lower extremities
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Patients: All study patients
Arm/Group | All Patients
Number analyzed (Participants) | 6
units on a scale | 4.5 (0.223)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: XTRAC excimer laser (wavelength of 308 nm) was performed using the standard vitiligo protocol of twice weekly treatments for twelve weeks. Standard safety vitiligo protocols were followed; for instance, if burning occurred, fluence was adjusted appropriately.
Arm/Group | Excimer Light Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Limitations included a small sample size with minimal variation in Fitzpatrick skin type, an all-female pool, and lack of extended follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No